CLINICAL TRIAL: NCT06448260
Title: Outcome of a Cohort of Patients Fitted With a SYME Type Prosthesis in the Context of a Hindfoot Amputation With Distal Support
Acronym: DEVSYME
Status: Completed | Type: Observational
Sponsor: Institut Robert Merle d'aubigné (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A00393-44
Record Dates: First submitted 2024-06-01; First posted 2024-06-07 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-10

CONDITIONS: Amputation, Surgical; Walking, Difficulty
Keywords: Amputation; Prothesis; Outcome
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with ATCT: Patient with tibiocalcaneal arthrodesis with talectomy amputation
  Interventions: Other: Questionnary

INTERVENTIONS:
Other: Questionnary — Data from theses patients will be collected in our personnal data base with ask of consent according to the law Then each patient alive will have questionnary to answer by phone or during a visit.

SUMMARY:
The purpose of this study is to see outcome of patients with syme prothesis in order to comment the handfoot amputation.

ELIGIBILITY:
Inclusion Criteria:

* Syme or Pirogoff or ATCT or arthrodesized Chopart type amputation
* Age > 18 years old,
* First fitting or renewal of Syme type prosthesis delivered to IRMA between January 2008 and December 2018

Exclusion Criteria:

* Refusal documented in the file that the data be used for scientific purposes,
* Congenital etiology of the condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient treated at the institut Rober Merle d'Aubigné
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The possibility of walking without a prosthesis | Immediatly after inclusion
  Yes / No
Walking perimeter with prosthesis | Immediatly after inclusion
  In meters
Number of re-amputation since first amputation | Immediatly after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Robert Merle d'Aubigné, Valenton, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Braaksma R, Dijkstra PU, Geertzen JHB. Syme Amputation: A Systematic Review. Foot Ankle Int. 2018 Mar;39(3):284-291. doi: 10.1177/1071100717745313. Epub 2018 Jan 10. PMID 29320640
- [Background] Dillon MP, Quigley M, Fatone S. Outcomes of dysvascular partial foot amputation and how these compare to transtibial amputation: a systematic review for the development of shared decision-making resources. Syst Rev. 2017 Mar 14;6(1):54. doi: 10.1186/s13643-017-0433-7. PMID 28288686
- [Background] van der Wal GE, Dijkstra PU, Geertzen JHB. Lisfranc and Chopart amputation: A systematic review. Medicine (Baltimore). 2023 Mar 10;102(10):e33188. doi: 10.1097/MD.0000000000033188. PMID 36897730
- [Background] Spoden M, Nimptsch U, Mansky T. Amputation rates of the lower limb by amputation level - observational study using German national hospital discharge data from 2005 to 2015. BMC Health Serv Res. 2019 Jan 6;19(1):8. doi: 10.1186/s12913-018-3759-5. PMID 30612550